CLINICAL TRIAL: NCT04271618
Title: Modulation of Sagittal Spinal Geometry in Children With Cerebral Palsy: Randomized Controlled Trial
Brief Title: Modulation of Sagittal Spinal Geometry in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Shamekh Mohamed El-Shamy, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Umm Al-Qura U
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Treatment Arm (Active Comparator): Participants in this group will receive conventional rehabilitation program for postural correction 2 hours/3 sessions' weekly/3 successive months.
  Interventions: Other: TheraTogs Orthotic Undergarment
- TheraTogs Undergarment Arm (Experimental): Participants in this group will receive the same conventional rehabilitation program as in traditional group in addition to wearing of TheraTogs soft orthotic undergarment with strapping system.
  Interventions: Other: TheraTogs Orthotic Undergarment

INTERVENTIONS:
Other: TheraTogs Orthotic Undergarment — Strapping undergarment made from a lightweight, breathable fabric that is velcro sensitive. It consists of sleeveless vest (tank-Top), two shorts (Hipster) each with two thigh cuffs and limb cuffs

SUMMARY:
The aim of this study will be to evaluate the the effect of Thera Togs soft orthotic undergarment on modulation of the spinal geometry and mobility in sagittal plan in children with spastic diplegic cerebral palsy.

DETAILED DESCRIPTION:
Forty children with spastic diplegic CP will be assigned and randomly distributed into two equall groups (A& B). Control group (A) will receive conventional rehabilitation program for postural correction 2 hours/3 sessions' weekly/3 successive months. Study group (B) will receive conventional rehabilitation protocol as in group (A) plus wearing TheraTogs soft orthotic undergarment. Children evaluation will be carried out before and after the intervention programs to assess postural deviations using the Formetric system.

ELIGIBILITY:
Inclusion Criteria:

* Have a definite diagnosis of spastic diplegia obtained from medical files or personal physicians and supported by magnetic resonance images (MRIs).
* Their weight should be less than 40 kg.
* The degree of spasticity in the affected lower extremity will ranged between grades (1, 1+&2) according to Modified Ashworth Scale.
* The levels of gross motor function will be selected at level II according to Gross Motor Function Classification System.
* The children will be included have the ability to stand alone for five minutes.
* Children should be able to understand and follow instructions.
* The degree of the spinal kyphosis ,for all participated children , in sagittal plane should be not more than 55° as Kyphosis above 55° is considered as fixed hyper-kyphosis while

Exclusion Criteria:

* Children with GMFCS levels III, IV, and V or use any assistive mobility devices
* Children suffering from allergic problems in their skin.
* Children with visual, auditory or cognitive deficits.
* Fixed and significant deformities of the lower limb and spine.
* Children with surgical interference for the lower limb and spine within the previous 2 years.
* Children with seizures.
* Children with fixed hyper-kyphosis (kyphotic angle is more than 55°).
* Children who used any medications (e.g., steroids) that affect growth or body composition.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Thoracic kyphotic angle at 3 months | Baseline and 3 months post-intervention
  Thoracic kyphotic angle will be calculated from the sagittal profile by Foremetric system.
Change from baseline lumber lordotic angle at 3 months | Baseline and 3 months post-intervention
  Lumber lordotic angle will be calculated from the sagittal profile by Foremetric system.

CONTACTS AND LOCATIONS:
Overall Officials: Shamekh M El-Shamy, Ph.D., Principal Investigator — Professor
Locations (1):
- Maternity and Children Hospital, Mecca, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No